CLINICAL TRIAL: NCT04021758
Title: Peer to Peer Programs for Military Suicide Prevention
Acronym: P2P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Xcelerate Innovations (Unknown)
Responsible Party: Principal Investigator, Craig Bryan, Associate Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PT170195; W81XWH-18-2-0064 (Other Grant/Funding Number: Congressionally Directed Medical Research Programs, USAMRMC)
Record Dates: First submitted 2019-05-02; First posted 2019-07-16 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Suicide
Keywords: Suicide prevention; Peer mentoring
MeSH Terms: conditions — Suicide; Suicide Prevention

STUDY DESIGN:
Intervention Model Description: The study design entails a dynamic wait list design in which participants are randomly assigned to either the Peer-to-Peer (P2P) program or a wait list control condition. Randomization will be conducted at the squadron level using a computerized randomization algorithm.
  The proposed dynamic wait list design differs primarily from the traditional wait list designs with respect to timing of intervention. In the traditional wait list design, half of the squadrons (i.e., N/2) would be randomized to implement the P2P program early in the study and the remaining half would implement the P2P program later in the study. By contrast, the dynamic wait list randomizes the timing of the intervention over the entire course of the study period by first dividing the overall study period into m equal time blocks, and then randomizing N/m squadrons to receive the P2P program during each time block.
Who Masked: Outcomes Assessor
Masking Description: Data analyses will be conducted by a quantitative psychology postdoctoral fellow under the supervision of Dr. Brian Baucom, PhD, at The University of Utah, and Kent Corso, PsyD, BCBA-D, at Xcelerate Innovations. Dr. Baucom serves on the University of Utah's Department of Psychology's Statistical Consulting Service, and has prior experience with clinical trial methodology and military research. Dr. Corso is a certified behavior analyst with extensive experience using single case design methodology and applying this approach to military settings. None of the data analysts will be involved in data collection procedures, and will remain therefore blind to treatment assignment. Prior to statistical analyses, data will be screened to identify distributional properties.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer to peer program intervention (Experimental): The experimental condition for the proposed project is the Airman's Edge program, a peer to peer program in which peer mentors will be trained to provide a series of interventions aimed at reducing risk for suicidal behaviors both directly and indirectly through the targeting of emotion dysregulation, cognitive rigidity, and contextual risk factors (e.g., insomnia, meaning in life, social support, firearm availability).
  Interventions: Behavioral: Peer to peer program intervention
- Wait list (No Intervention)

INTERVENTIONS:
Behavioral: Peer to peer program intervention — Peer to peer suicide prevention program aimed at reducing suicide in a military population.
  Other Names: Airman's Edge
  Arms: Peer to peer program intervention

SUMMARY:
In the present project the investigators propose to test the efficacy of a peer to peer program entitled Airman's Edge. The Airman's Edge program plans to utilize peer mentors that will be trained in specialized skills designed to impact suicide risk at multiple levels of the military community without creating "extra duties" that increase workload and interfere with mission demands. Peer mentors will introduce primary prevention strategies to their units that target broad-based risk factors across the entire population (i.e., sleep disturbance, social support, meaning in life, firearm safety) with secondary prevention strategies that target individual-level risk factors (i.e., crisis response planning, firearm safety counseling). Peer mentors will complete a structured training process using existing curriculum and procedures that have been tested and refined within military groups. Peers mentors will also participate in monthly consultation calls with the investigative team to receive ongoing support, share resources and lessons learned, and address challenges and barriers to program implementation.

The purpose of the Airman's Edge peer to peer program is to influence indicators of suicide risk among military personnel at two levels, group and individual, consistent with the program's hybrid design that combines group-based education and individual-level suicide prevention skills training. The hypotheses are therefore designed to examine outcomes and effects at multiple levels of the community, which could inform subsequent implementation and translational efforts. The following aims are proposed:

Aim 1: To test the efficacy of a peer to peer program for the reduction of suicidal behavior among military personnel.

Aim 2: To identify moderators and mediators of the peer to peer program's effects on suicidal behavior.

DETAILED DESCRIPTION:
Suicides among military personnel doubled from 2001 to 2015 and have remained elevated. Although new treatments and interventions have been shown to reduce the occurrence of suicidal behavior, they are predominantly available only in mental health clinics. Data indicates that the large majority of military personnel who die by suicide do not access mental healthcare services in the months preceding their deaths. New strategies that are based on these empirically-supported interventions but can be delivered outside the mental healthcare system, thereby reaching a larger proportion of the military community, are therefore needed. Peer to peer (P2P) support programs hold promise as a method for achieving these aims, but the evidence supporting this intervention model remains limited or, in the case of suicide prevention, absent. In light of this gap, the proposed project aims to test the efficacy of a P2P program for the reduction of suicidal behaviors among military personnel. The proposed P2P program, called Airman's Edge, is a hybrid model that includes both group-based peer educator and individual-based peer support components; these P2P program models have demonstrated the strongest outcomes with respect to changing attitudes, perspectives, and behaviors, all of which are key targets for reducing suicidal thoughts and behaviors. The Airman's Edge program is comprised of several skills-based strategies that have been shown to directly reduce suicidal thoughts and behaviors (i.e., sleep habits, firearm safety procedures, crisis response planning), and targets population-level contextual variables known to reduce suicide risk (i.e., purpose and meaning in life, social support). The mechanisms by which these strategies reduce suicidal behavior align with an empirically-supported conceptual model, the suicidal mode, which has guided recent advances in military suicide prevention. The delivery platform for the skills-based strategies employed in the Airman's Edge program have demonstrated very good acceptability and feasibility when used with military personnel.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older; and
2. able to understand and speak the English language.

Exclusion Criteria:

1. an inability to understand and speak the English language and
2. an inability to complete the informed consent process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2055 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Change in number of suicide deaths from baseline | Administrative data will be requested at baseline for the five years preceding the start of the study, and will be requested on a quarterly basis through study completion, an average of 20 months.
  Number of suicide deaths will be collected from Department of Defense Suicide Event Report data.
Change in suicidal behaviors from baseline | Participants will complete self-report assessments at baseline and every four months during follow-up for a total of 20 months.
  Include suicide attempts, aborted suicide attempts, and interrupted suicide attempts. Will be assessed using the self-report version of the Self-Injurious Thoughts and Behaviors Interview (SITBI; Nock et al., 2007). The SITBI is a PhenX Toolkit recommended common data element.
Change in suicide ideation from baseline | . Participants will complete self-report assessments at baseline and every four months during follow-up for a total of 20 months.
  Suicide ideation will be assessed using the self-report version of the Self-Injurious Thoughts and Behaviors Interview (SITBI; Nock et al., 2007). The SITBI is a PhenX Toolkit recommended common data element.

CONTACTS AND LOCATIONS:
Overall Officials: Craig J Bryan, PsyD, Principal Investigator — The University of Utah
Locations (1):
- Whiteman Air Force Base, Whiteman Air Force Base, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bryan, C. J., & Morrow, C. E. (2011). Circumventing mental health stigma by embracing the warrior culture: Lessons learned from the Defender's Edge program. Professional Psychology: Research and Practice, 42(1), 16-23. https://doi.org/10.1037/a0022290
- [Background] Bryan CJ, Mintz J, Clemans TA, Burch TS, Leeson B, Williams S, Rudd MD. Effect of Crisis Response Planning on Patient Mood and Clinician Decision Making: A Clinical Trial With Suicidal U.S. Soldiers. Psychiatr Serv. 2018 Jan 1;69(1):108-111. doi: 10.1176/appi.ps.201700157. Epub 2017 Oct 2. PMID 28967323
- [Background] Bryan CJ, Mintz J, Clemans TA, Leeson B, Burch TS, Williams SR, Maney E, Rudd MD. Effect of crisis response planning vs. contracts for safety on suicide risk in U.S. Army Soldiers: A randomized clinical trial. J Affect Disord. 2017 Apr 1;212:64-72. doi: 10.1016/j.jad.2017.01.028. Epub 2017 Jan 23. PMID 28142085
- [Background] Bryan CJ, Andreski SR, McNaughton-Cassill M, Osman A. Agency is associated with decreased emotional distress and suicidal ideation in military personnel. Arch Suicide Res. 2014;18(3):241-50. doi: 10.1080/13811118.2013.824836. PMID 24712868
- See also: National Center for Veterans Studies — https://veterans.utah.edu/